CLINICAL TRIAL: NCT01001364
Title: A Phase III, Randomized, Open-Label, Non-Inferiority Comparative Study Between Foraseq Inhalation Capsules 12/200 Μg and Formoterol/ Budesonide Inhalation Capsules 12/200 Μg Eurofarma in Patients with Asthma
Brief Title: A Comparative Study Between Foraseq and Formoterol/Budesonide Inhalation Capsules in Patients with Asthma
Acronym: CAINAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-091
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: ASTHMA
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Formoterol/Budesonide (Experimental)
  Interventions: Drug: Formoterol/Budesonide
- Foraseq (Active Comparator)
  Interventions: Drug: Foraseq

INTERVENTIONS:
Drug: Formoterol/Budesonide — formoterol will be administered at the 12 µg dosage, twice a day, and budesonide will be administered at the 200 µg dose, also twice a day for 12 weeks.
  Arms: Formoterol/Budesonide
Drug: Foraseq — formoterol will be administered at the 12 µg dosage, twice a day, and budesonide will be administered at the 200 µg dose, also twice a day for 12 weeks.
  Arms: Foraseq

SUMMARY:
This study primary objective is to compare the impact of two products containing budesonide and formoterol as individual capsules with inhalation powder for the pulmonary function of subjects with persistent asthma.

DETAILED DESCRIPTION:
This study primary objective is to compare the impact of two products containing budesonide and formoterol as individual capsules with inhalation powder for the pulmonary function of subjects with persistent asthma. This is a non-inferiority study, which hypothesis is that there is no difference on the pulmonary function measure between the groups studied at its end. Therefore, the study primary endpoint will be the forced expiratory volume in 1 second (FEV1) at the final visit (FV) at each study arm.

This study secondary objective is to compare the impact on the clinical control of two products containing budesonide and formoterol as individual capsules with inhalation powder in subjects with persistent asthma.

The secondary endpoints considered for this study are:

* Score of asthma control questionnaire (ACQ-7) 34 at the end of the study ;
* Peak of expiratory flow (PEF) throughout the study;
* Symptoms score at the end of the study;
* FEV1 throughout the study;
* Treatment safety, including serum cortisol dosage;
* Frequency of observed adverse events.

Some eligibility criteria:

* Current use of inhaled corticosteroids (equivalent to beclometasone dipropionate 1000µg) associated or not to long-acting β2-adrenergics and relief medication (salbutamol or equivalent);
* Diagnosis of mild to moderate persistent asthma, as per the ARIA classification, 35 with symptoms for at least 6 months, clinically stable for at least 1 month with ACQ-7 test34 (see Attachment D) < 3.0;

ELIGIBILITY:
Inclusion Criteria:

* Sign ICF (see Attachment A);
* Age ≥12 years old
* Diagnosis of mild to moderate persistent asthma, as per the ARIA classification, 35 with symptoms for at least 6 months, clinically stable for at least 1 month with ACQ-7 test34 (see Attachment D) < 3.0;
* Current use of inhaled corticosteroids (equivalent to beclometasone dipropionate 1000µg) associated or not to long-acting β2-adrenergics and relief medication (salbutamol or equivalent);
* Initial FEV1 of at least 50% of the normal value estimated.
* Serum cortisol evaluation within the normal values

Exclusion Criteria:

* Use of oral or parenteral corticosteroids within the last 3 months;
* Need of hospitalization due to asthma within the last 3 months;
* Active tabagism, defined as the use of cigarettes, pipe, cigar or any other type in any amount within the last 3 months;
* Severe co-morbidity, such as cardiovascular, renal, liver, neurologic, neoplastic, blood, infectious, dermatologic, neurologic, psychiatric or chronic respiratory diseases, other than asthma;
* Recent participation (<6 months) or planned participation, during this study, on other clinical trials involving drugs of any nature or under studies of any type of intervention for the asthma treatment;
* Intolerance or allergy to any of the compounds of the drugs evaluated on the study;
* Pregnancy or lactation;
* Chronic use of routine oral or intravenous β-blocker drugs, even ophthalmic solutions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The study primary endpoint will be the forced expiratory volume in 1 second (FEV1) at the final visit (FV) at each study arm. | 4 months

SECONDARY OUTCOMES:
Only one Score of asthma control questionnaire (ACQ-7) 34 at the end of the study. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Pesquisa Clínica Stelmach, São Paulo, São Paulo, Brazil